CLINICAL TRIAL: NCT01151345
Title: Bioequivalence Study Of Diltiazem In 60 Mg Tablets As Tilazem 60® Made By Pfizer, S.A. DE C.V., Versus Angiotrofin® 60 Mg Made By Amstrong Laboratorios De Mexico, S.A. DE C.V. Study In 26 Healthy Volunteers Of Both Genders Under Fasting Conditions
Brief Title: Bioequivalence Study Of Diltiazem In 60 Mg Tablets As Tilazem 60® Made by Pfizer, S.A. De C.V., Versus Angiotrofin® 60 Mg Made by Amstrong Laboratorios De Mexico, S.A. De C.V.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A7661002
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Results first posted 2011-08-22 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: diltiazem; angiotrofin; bioequivalence
MeSH Terms: interventions — angiotrofin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diltiazem (Experimental)
  Interventions: Drug: TILACEM; Drug: ANGIOTROFIN

INTERVENTIONS:
Drug: TILACEM — At 08:00 hours on day 1, CIF-BIOTEC personnel will start to administer the study drug. Each volunteer will receive a single dose of 60 mg of Diltiazem. The study drugs will be ingested with 250 mL of drinking water. Research Pharmacy personnel will inspect the volunteer's oropharynx to ensure that he/she has swallowed the tablet and record their observations in the corresponding forms.
Drug: ANGIOTROFIN — At 08:00 hours on day 1, CIF-BIOTEC Pharmacy personnel will start to administer the study drug. Each volunteer will receive a single dose of 60 mg of Diltiazem. The study drugs will be ingested with 250 mL of drinking water. Research Pharmacy personnel will inspect the volunteer's oropharynx to ensure that he/she has swallowed the tablet and record their observations in the corresponding forms.

SUMMARY:
This study will research the existance of actual bioequivalence between Diltiazem in 60 Mg Tablets As Tilazem 60® Made by Pfizer, S.A. DE C.V., Versus Angiotrofin® 60 Mg Made by Amstrong Laboratorios De Mexico, S.A. DE C.V.

DETAILED DESCRIPTION:
Bioequivalence of this particular drug

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Both genders
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2 or ± 10% variation of the ideal weight; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Mexico City, Mexico City, Mexico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7661002&StudyName=Bioequivalence%20Study%20Of%20Diltiazem%20In%2060%20Mg%20Tablets%20As%20Tilazem%2060%AE%20Made%20by%20Pfizer%2C%20S.a.%20De%20C.v.%2C%20Versus%20Angiotrofin%AE%2060%20Mg%20Ma

RESULTS

PARTICIPANT FLOW:
Groups:
- Tilazem 60 mg Then Angiotrofin 60 mg: Single oral dose of 60 mg Diltiazem tablet (Tilazem®) in first intervention period and single oral dose of 60 mg Diltiazem tablet (Angiotrofin®) in second intervention period after 7 day clearance period. The total study duration was 9 days.
- Angiotrofin 60 mg Then Tilazem 60 mg: Single oral dose of 60 mg Diltiazem tablet (Angiotrofin®) in first intervention period and single oral dose of 60 mg Diltiazem tablet (Tilazem®) in second intervention period after 7 day clearance period.The total study duration was 9 days.
Period: First Intervention Period
Arm/Group | Tilazem 60 mg Then Angiotrofin 60 mg | Angiotrofin 60 mg Then Tilazem 60 mg
Started | 13 | 13
Treated | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Wash-out Period (7 Days)
Arm/Group | Tilazem 60 mg Then Angiotrofin 60 mg | Angiotrofin 60 mg Then Tilazem 60 mg
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | Tilazem 60 mg Then Angiotrofin 60 mg | Angiotrofin 60 mg Then Tilazem 60 mg
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive any treatment (Tilazem 60 mg tablet first or Angiotrofin 60 mg tablet first )
Arm/Group | Entire Study Population
Number analyzed (Participants) | 26
Age Continuous [Mean (Standard Deviation); unit: Years] | 33.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)]
Description: AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post dose
Population: Pharmacokinetic (PK) parameter analysis population included all treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Tilazem 60 mg: Single oral dose of 60 mg Diltiazem tablet (Tilazem®) in either first intervention period or second intervention period.
- Angiotrofin 60 mg: Single oral dose of 60 mg Diltiazem tablet (Angiotrofin®) in either first intervention period or second intervention period.
Arm/Group | Tilazem 60 mg | Angiotrofin 60 mg
Number analyzed (Participants) | 25 | 25
ng*hr/mL | 463.41 (245.03) | 498.87 (226.07)
Statistical Analysis 1: Comparison: Tilazem 60 mg vs Angiotrofin 60 mg; Natural-log transformed AUC (0-t) was analyzed using a mixed effect model with sequence, period, and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Adjusted geometric means ratio = 88.65, 90% CI 2-sided [81.23 to 96.75]

2. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)]
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Tilazem 60 mg | Angiotrofin 60 mg
Number analyzed (Participants) | 25 | 25
ng*hr/mL | 612.95 (298.23) | 648.68 (283.73)
Statistical Analysis 1: Comparison: Tilazem 60 mg vs Angiotrofin 60 mg; Natural-log transformed AUC (0-∞) was analyzed using a mixed effect model with sequence, period, and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Adjusted geometric means ratio = 91.26, 90% CI 2-sided [83.83 to 99.34]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post dose
Population: PK parameter analysis population included all treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tilazem 60 mg | Angiotrofin 60 mg
Number analyzed (Participants) | 25 | 25
ng/mL | 68.67 (50.36) | 79.60 (44.01)
Statistical Analysis 1: Comparison: Tilazem 60 mg vs Angiotrofin 60 mg; Natural-log transformed Cmax was analyzed using a mixed effect model with sequence, period, and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; Adjusted geometric means ratio = 83.25, 90% CI 2-sided [67.08 to 103.31]

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Tilazem 60 mg | Angiotrofin 60 mg
Number analyzed (Participants) | 25 | 25
hr | 2.38 (0.98) | 2.44 (1.04)

5. Primary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 24 hours post dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Tilazem 60 mg | Angiotrofin 60 mg
Number analyzed (Participants) | 25 | 25
hr | 12.17 (5.98) | 11.71 (5.55)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tilazem 60 mg | Angiotrofin 60 mg
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 10/25 | 13/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tilazem 60 mg (N=25) | Angiotrofin 60 mg (N=25)
Headache (General disorders) | 5 | 6
Dizziness (General disorders) | 4 | 4
Diarrhoea (General disorders) | 1 | 2
Gastrointestinal pain (General disorders) | 1 | 0
Hypoaesthesia (General disorders) | 1 | 0
Muscular weakness (General disorders) | 1 | 0
Tremor (General disorders) | 1 | 0
Blepharitis (General disorders) | 0 | 1
Nausea (General disorders) | 0 | 1
Somnolence (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.